CLINICAL TRIAL: NCT03574506
Title: Eculizumab Use in the Postpartum Period for the Treatment of Pregnancy Associated Atypical Hemolytic Uremic Syndrome: A Case Series
Brief Title: Eculizumab Use in the Postpartum Period for the Treatment of Pregnancy Associated aHUS: A Case Series
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Grupo de Investigación en Cuidados Intensivos y Obstetricia (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LS30885-1
Record Dates: First submitted 2018-05-24; First posted 2018-07-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Atypical Hemolytic Uremic Syndrome; Pregnancy
Keywords: Atypical Hemolytic Uremic Syndrome; Pregnancy
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eculizumab is a humanized monoclonal IgG antibody against protein C5 that works to inhibit the activation of the terminal complement cascade. The Eculizumab is currently FDA approved for the treatment of Paroxysmal nocturnal hemoglobinuria and atypical hemolytic uremic syndrome (aHUS) and has been shown to improve the quality of life and overall survival in these patients. aHUS is a life-threatening disease of complement mediated thrombotic microangiopathy often triggered by an inciting event, such as an infection or immunocompromised state. Pregnancy has also been identified as an inciting event, with patients most often experiencing aHUS in the postpartum period. Due to its rare nature, pregnancy-associated aHUS is often mistaken for preeclampsia or hemolysis, elevated liver enzyme, low platelet (HELLP) syndrome. As standard treatment for preeclampsia and HELLP syndrome is completion of the pregnancy by expediting delivery of the baby. A missed diagnosis of aHUS can result in delays in treatment, including use of Eculizumab when appropriate; such delay can increase the risk of maternal morbidity and mortality. When aHUS is suspected in the postpartum period, Eculizumab could be initiated early; however, there is limited data on use of Eculizumab in this setting.

DETAILED DESCRIPTION:
Overall Objective The aim of this study is compare outcomes of women with suspected postpartum aHUS, stratified by treatment with Eculizumab. Specifically, assess the maternal characteristics, clinical presentation, disease course, treatment strategy, and short and long--term complications among a cohort of women with suspected postpartum aHUS, with analyses stratified by Eculizumab exposure.

Aim 1 Hypothesis: Women with suspected postpartum aHUS treated with Eculizumab have a decreased length of hospital stay and a decreased incidence of adverse maternal outcomes when compared to those women with postpartum aHUS not treated with Eculizumab.

Aim 2 Hypothesis: Women with postpartum aHUS treated with Eculizumab have low rates of adverse maternal or neonatal events when followed up to 6 months after delivery.

METHODOLOGY Study Type: Retrospective cohort study Study population: Postpartum patients meeting diagnostic criteria for pregnancy associated aHUS between January 2009 and May 2016 in Colombia. This study cohort will be stratified into two groups: 1) women with suspected postpartum aHUS treated with Eculizumab and; 2) women meeting diagnostic criteria for postpartum aHUS that did not receive treatment with Eculizumab. The investigators chose a start date of 2009 because this was the year that Eculizumab was approved by the National Institute of Food and Drug Monitoring (INVIMA) for use in Paroxysmal Nocturnal Hemoglobinuria (PNH). Eculizumab was subsequently approved for use in aHUS in 2011.In addition, in the same period of time will identify a cohort of women diagnosed with pregnancy associated with HUS in Colombia who did not receive treatment with Eculizumabse.

Unit of analysis: The medical data of patients who meet the inclusion criteria for the study, ie, postpartum aHUS are summarized. For the group of women treated with Eculizumab, and who continue to receive such therapy on an outpatient basis after hospital discharge, the investigators will abstract follow up data up to 6 months postpartum. For missing data that is not readily available in the medical chart the investigators will utilize research assistants, or members of the study team, to contact study subjects or the treating provider to obtain additional information.

Will be assessed sample size requirements necessary to determine a significant difference in survival or end--stage renal disease between groups (primary outcomes), with 80% power and alpha=0.05 (see tables below). Mortality from aHUS without Eculizumab in Colombia is estimated at 30% based in previous reports. The investigators estimate out treatment cohort of aHUS cases treated with Eculizumab to be at least Ten patients. Thus, the investigators have sufficient power to detect a significant increase in overall survival if it is 80% or greater in the treatment arm. Rate of end-stage renal disease (ESRD) with aHUS is estimated at 70% in Colombia. The investigators have sufficient to detect a significant decrease in ESRD with Eculizumab if the rate is 15% or lower.

The study will consist of three steps:

Step 1: Identification of study cohort Activity 1: This project will be submitted to Alexion Pharma SAS in Colombia, in order to obtain approval and access to information on all patients in their database who received treatment with Eculizumab after being diagnosed with postpartum aHUS regardless of outcome. Alexion is the only authorized distributor of Eculizumab by the National Institute of Food and Drug Monitoring (INVIMA).

Activity 2: Obtaining informed consent from all patients meeting criteria for postpartum aHUS, regardless of Eculizumab treatment, to access data from medical records or directly via interviews with study subjects or their representatives.

Activity 3: Written and verbal communication to the various medical providers involved in the care of the identified patient cohort. For this study, were defined as those providers who made the initial and / or final diagnosis of pregnancy associated aHUS and who were responsible for treatment of the patient.

Step 2: Review of information and data collection:

Activity 1: Review all information obtained from the medical records of all subjects meeting inclusion criteria by the investigators. A database will then be constructed and populated with the information obtained.

Activity 2: Data Verification A second researcher will conduct a verification of the information included in the database, to assess quality control of the data entered.

Stage 3: Analysis of results Activity 1: To describe clinical and sociodemographic characteristics, disease course, and treatment approach in patients with postpartum aHUS.

Activity 2: To assess adverse maternal outcomes among women with postpartum aHUS, stratified by treatment with Eculizumab. Short term outcomes will be assessed from the time of diagnosis to the time of hospital discharge.

Activity 3: To determine the rate of delayed adverse maternal and neonatal events in women with postpartum aHUS treated with Eculizumab, and who are followed up to 6 months after delivery.

The database in an excel spreadsheet format will be used to conduct descriptive analysis of the demographic variables and subject characteristics. Correlations of outcomes will be made with timing of initiation of Eculizumab after delivery, dose received.

Clinical variables Demographic characteristics, Obstetric history, Characteristics of current pregnancy Clinical criteria (At time of presentation, diagnosis, and after treatment) Laboratory test (if possible) (At presentation, diagnosis, and throughout treatment course) Treatments Eculizumab treatment Maternal outcomes Neonatal outcomes

ETHICAL CONSIDERATIONS Throughout the study period the investigators will ensure the confidentiality of information collected, the accuracy of the results obtained, and above all the investigators respect the ights of all patients involved. All copies of signed consent forms and medical records retrieved will be stored in a locked cabinet in the principal investigators office.

This research study is classified as "safe", according to Article 11 of resolution 8430 of 1993 by the Ministry of Health of Colombia.

The data collected during the study will be used solely for research purposes and all appropriate measures will be taken to keep information confidential. Prior to proceeding this project will be approved by the Ethic Committee of the hospital ESE Divina Misericordia from Magangué, Colombia (see attached in appendix the Spanish version in PDF format), and will be submitted to the institutional review board of Oregon Health & Science University.

This study fits within the ethical guidelines of the Helsinki statement and the ethical principles of the World Medical Association. As stated prior, all the information collected for this investigation will be confidential and the results will be published only in journals with academic and scientific interest, preserving the accuracy of the data as well as the findings and results.

Alexion Pharma SAS in Colombia will provide the information of patients who received Eculizumab for treatment of atypical hemolytic uremic syndrome in the postpartum period. After obtaining patient consent the investigators will then access their medical record information and ensure all information is collected in a secure database.

Alexion Pharma SAS in Colombia is the only authorized distributor of Eculizumab by the National Institute of Food and Drug Monitoring (INVIMA). Alexion Pharma SAS will receive a copy of the analysis and report which will be published in an independent manner by the investigators.

This protocol complies with the ethical requirements for human research outlined by the American Medical Association such as its scientific value, describing the impact generated using Eculizumab, a monoclonal antibody, on the natural history and progression of aHUS during pregnancy and/or the postpartum period and therefore, to raise future clinical research in terms of reduction of morbidity and mortality related to this disease.

Finally, only patients who have given their informed consent will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the postpartum period (within 12 weeks of delivery) that were diagnosed with aHUS by their treating provider or who met standard diagnostic criteria.
* Subjects meeting diagnostic criteria for aHUS will be included in the study independent of the treatment approach employed by their providers.
* Those who received at least one dose of Eculizumab for treatment of suspected aHUS will be included, regardless of outcome.

Exclusion Criteria:

* Patients who did not authorize the use of their information after an informed consent process
* Patients who their physicians who did not agree to participate in or provide patient information.

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Postpartum patients meeting diagnostic criteria for pregnancy associated aHUS between January 2009 and May 2016 in Colombia. This study cohort will be stratified into two groups: 1) women with suspected postpartum aHUS treated with Eculizumab and; 2) women meeting diagnostic criteria for postpartum aHUS that did not receive treatment with Eculizumab. We chose a start date of 2009 because this was the year that Eculizumab was approved by the National Institute of Food and Drug Monitoring (INVIMA) for use in Paroxysmal Nocturnal Hemoglobinuria (PNH). Eculizumab was subsequently approved for use in aHUS in 2011. We also seek to identify a matched cohort of women diagnosed with pregnancy associated aHUS in Colombia in the same time frame who did not receive Eculizumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Maternal mortality | The data collection will be among the first postpartum day until the sixth month
  Death of a woman within 42 days of termination of pregnancy. This is a dichotomy measure

SECONDARY OUTCOMES:
ICU length of stay | The data collection will be among the first postpartum day until the sixth month
  Time (in days) of stay in an intensive care unit from admission to discharge or death of the patient. This is a continuous measure
Dosing and number of doses received | The data collection will be among the first postpartum day until the sixth month
  Dosage of eculizumab (in mg) per day received by the woman with a diagnosis of atypical hemolytic uremic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rojas, MD. Msc, Principal Investigator — Fundacion GRICIO
Locations (1):
- Gestion Salud, Cartagena, Departamento de Bolívar, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noris M, Remuzzi G. Atypical hemolytic-uremic syndrome. N Engl J Med. 2009 Oct 22;361(17):1676-87. doi: 10.1056/NEJMra0902814. No abstract available. PMID 19846853
- [Background] Fakhouri F, Hourmant M, Campistol JM, Cataland SR, Espinosa M, Gaber AO, Menne J, Minetti EE, Provot F, Rondeau E, Ruggenenti P, Weekers LE, Ogawa M, Bedrosian CL, Legendre CM. Terminal Complement Inhibitor Eculizumab in Adult Patients With Atypical Hemolytic Uremic Syndrome: A Single-Arm, Open-Label Trial. Am J Kidney Dis. 2016 Jul;68(1):84-93. doi: 10.1053/j.ajkd.2015.12.034. Epub 2016 Mar 21. PMID 27012908
- [Background] Kelly RJ, Hochsmann B, Szer J, Kulasekararaj A, de Guibert S, Roth A, Weitz IC, Armstrong E, Risitano AM, Patriquin CJ, Terriou L, Muus P, Hill A, Turner MP, Schrezenmeier H, Peffault de Latour R. Eculizumab in Pregnant Patients with Paroxysmal Nocturnal Hemoglobinuria. N Engl J Med. 2015 Sep 10;373(11):1032-9. doi: 10.1056/NEJMoa1502950. PMID 26352814
- [Background] Kelly RJ, Hill A, Arnold LM, Brooksbank GL, Richards SJ, Cullen M, Mitchell LD, Cohen DR, Gregory WM, Hillmen P. Long-term treatment with eculizumab in paroxysmal nocturnal hemoglobinuria: sustained efficacy and improved survival. Blood. 2011 Jun 23;117(25):6786-92. doi: 10.1182/blood-2011-02-333997. Epub 2011 Apr 1. PMID 21460245
- [Background] Fakhouri F, Roumenina L, Provot F, Sallee M, Caillard S, Couzi L, Essig M, Ribes D, Dragon-Durey MA, Bridoux F, Rondeau E, Fremeaux-Bacchi V. Pregnancy-associated hemolytic uremic syndrome revisited in the era of complement gene mutations. J Am Soc Nephrol. 2010 May;21(5):859-67. doi: 10.1681/ASN.2009070706. Epub 2010 Mar 4. PMID 20203157
- [Background] Tsai HM, Kuo E. From Gestational Hypertension and Preeclampsia to Atypical Hemolytic Uremic Syndrome. Obstet Gynecol. 2016 May;127(5):907-910. doi: 10.1097/AOG.0000000000001340. PMID 27054930
- [Background] Vaught AJ, Gavriilaki E, Hueppchen N, Blakemore K, Yuan X, Seifert SM, York S, Brodsky RA. Direct evidence of complement activation in HELLP syndrome: A link to atypical hemolytic uremic syndrome. Exp Hematol. 2016 May;44(5):390-8. doi: 10.1016/j.exphem.2016.01.005. Epub 2016 Feb 26. PMID 26921648
- [Background] Emanuel EJ, Wendler D, Grady C. What makes clinical research ethical? JAMA. 2000 May 24-31;283(20):2701-11. doi: 10.1001/jama.283.20.2701. PMID 10819955